CLINICAL TRIAL: NCT04263402
Title: An Open, Prospective/Retrospective, Randomized Controlled Cohort Study to Compare the Efficacy of Different Hormone Doses in the Treatment of 2019-nCoV Severe Pneumonia
Brief Title: The Efficacy of Different Hormone Doses in 2019-nCoV Severe Pneumonia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Qin Ning, Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TJ20200201
Record Dates: First submitted 2020-02-02; First posted 2020-02-10 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: 2019-nCoV Severe Pneumonia
MeSH Terms: interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methylprednisolone(<40mg/d) (Experimental)
  Interventions: Drug: Methylprednisolone
- Methylprednisolone(40~80mg/d) (Experimental)
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Methylprednisolone — Patients in the Group I will receive basic symptomatic supportive treatment,plus methylprednisolone(<40mg/d intravenous drip for 7 days).
  Arms: Methylprednisolone(<40mg/d)
Drug: Methylprednisolone — Patients in the Group II will receive basic symptomatic supportive treatment,plus methylprednisolone(40~80mg/d intravenous drip for 7 days).
  Arms: Methylprednisolone(40~80mg/d)

SUMMARY:
At present, there is no specific and effective antiviral therapy.In this study, an open, prospective/retrospective, randomized controlled cohort study was designed to compare the efficacy of different hormone doses in the treatment of 2019-nCoV severe Pneumonia.This study explores effective treatment programs for 2019-nCoV severe pneumonia and provides a reliable evidence-based basis for the treatment.

ELIGIBILITY:
Inclusion Criteria:

1.Meet the definition of severe pneumonia(Comply with any of the followings):

1. Shortness of breath,RR≥30 bpm;
2. In a resting state:SPO2≤93%;
3. PaO2/FiO2≤300mmHg.

2.2019-nCoV nucleic acid test was positive.

3.CT of the lung conformed to the manifestation of viral pneumonia.

Exclusion Criteria:

1. dying state (i.e. survival time is less than 24 hours);
2. progressive malignant tumor with life expectancy less than 6 months;
3. immunosuppressive status(patients using immunosuppressants or chemotherapeutic drugs)
4. underlying diseases requiring long-term glucocorticoid treatment in the past 6 months or short-term glucocorticoid therapy in the past 4 weeks;
5. pregnancy
6. patients with glucocorticoid taboos

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Rate of disease remission | day 7
  For mild patients: disease remission refers to relieved symptoms with improved lung CT; For severe patients: disease remission refers to relieved symptoms with improved lung CT; or SPO2>93% or PaO2/FiO2 >300mmHg.
Rate and time of entering the critical stage | day 7
  the critical stage refers to respiratory failure that occurs and requires mechanical ventilation, shock, or having other organ failure that needs ICU monitoring and treatment.

SECONDARY OUTCOMES:
Rate of normal tempreture | day 7
  Rate of patients without fever at day 7
Rate of respiratory symptom remission | day 7
  Rate of patients with respiratory symptom remission at day 7
Rate of lung imaging recovery | day 7
  Rate of patients with lung imaging recovery at day 7
Rate of laboratory indicator recovery | day 7
  Rate of patients with laboratory indicator recovery at day 7
Rate of undetectable viral RNA | day 7
  Rate of patients withundetectable viral RNA at day 7

CONTACTS AND LOCATIONS:
Locations (1):
- Department and Institute of Infectious Disease, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided